CLINICAL TRIAL: NCT04826068
Title: The Application and Modification of an Emotional Processing Intervention for Children With Traumatic Brain Injury
Brief Title: Emotional Processing Intervention for Children With TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Jean Lengenfelder, Assistant Director, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-11220-20
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Traumatic Brain Injury
Keywords: Emotional Processing; Pediatric Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Processing (Experimental): The intervention looks at emotional processing of face interpretation.
  Interventions: Behavioral: Emotional Processing
- Control intervention (Placebo Comparator): The control group is seeing the same faces and are asked questions regarding them.
  Interventions: Behavioral: Emotional Processing

INTERVENTIONS:
Behavioral: Emotional Processing — Processing Emotions of others based on photographs of faces

SUMMARY:
Investigating an emotional processing program, that is modified for use with children, is effective for children with a traumatic brain injury (TBI).

DETAILED DESCRIPTION:
The first stage of this project will evaluate the appropriateness of an emotional processing intervention modified for a pediatric population. The researchers will modify the intervention prior to the evaluation by the 15 typically developing children.

The second stage of the project will evaluate the effectiveness of an emotional processing intervention to improve performance on tests of emotional processing in individuals with TBI. Emotional processing includes both facial affect recognition and social perception measures.

ELIGIBILITY:
Inclusion Criteria:

Ages of 9 and 17. Speak and read English fluently.

Healthy Volunteer or

Have sustained a TBI at least 1 year ago, that has affected his or her ability to process emotions.

Exclusion Criteria:

Previous stroke, MS, or neurological injury or disease in the past (like brain tumor or epilepsy) other than TBI.

History of significant psychiatric illness (like bipolar disorder, schizophrenia or psychosis).

Uncontrolled seizures or other unstable medical complications.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Facial Identification Task | 8 weeks
  measure of facial affect recognition

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kessler Foundation, East Hanover, New Jersey
  - Kessler Foundation, West Orange, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided